CLINICAL TRIAL: NCT03173014
Title: EEG Finding in Moyamoya Disease in Children
Brief Title: EEG Monitoring in Children With Moyamoya Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, MD, PhD, Professor, Seoul National University Hospital
Other Study IDs: 1705-013-851
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: EEG With Periodic Abnormalities
MeSH Terms: interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: EEG — EEG monitoring

SUMMARY:
EEG in moyamoya disease in children preoperatively

DETAILED DESCRIPTION:
EEG monitoring in children with moyamoy disease preoperatively for 10 minutes

ELIGIBILITY:
Inclusion Criteria:

* moyamoya disease

Exclusion Criteria:

* refusal

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with moyamoya disease from 5-10 years old
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-05-30 (Estimated); Study Completion 2018-06-05 (Estimated)

PRIMARY OUTCOMES:
EEG | preoperative
  EEG finding

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, Principal Investigator — Seoul National University Children's Hospital
Locations (2):
- South Korea (2):
  - Hee-Soo Kim, Seoul, Soul-t'ukpyolsi
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided